CLINICAL TRIAL: NCT06191133
Title: Window of Opportunity Trial of Fenofibrate in Patients With High-grade Cervical Intraepithelial Neoplasia and Invasive Cervical Carcinoma
Brief Title: Fenofibrate in Patients With Cervical Intraepithelial Neoplasia and Invasive Cervical Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lindsay Ferguson, MD (Other)
Responsible Party: Sponsor-Investigator, Lindsay Ferguson, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE3822
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cervical Intraepithelial Neoplasia; Invasive Cervical Cancer
Keywords: Fenofibrate
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Fenofibrate; Conization; Hysterectomy; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Excisional procedure + Fenofibrate (Experimental): Participants with high-grade dysplasia will receive 200mg of Fenofibrate starting on the day of enrollment and will continue the drug administration daily for 2-4 weeks +/- 7 days until their excisional procedure
  Interventions: Drug: Fenofibrate; Procedure: Cervical Conization
- Hysterectomy or chemoradiation + fenofibrate (Experimental): Participants with invasive cervical cancer will receive 200mg of Fenofibrate starting on the day of enrollment and will continue the drug administration daily for 2-4 weeks +/- 7 days until their definitive hysterectomy or chemoradiation
  Interventions: Drug: Fenofibrate; Procedure: Hysterectomy; Radiation: Chemoradiation

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate is an FDA approved drug for cardiovascular indications and have decades of data supporting a favorable safety profile event with chronic use.
  Other Names: Antara; Fenoglide; Lipofen; Tricor; Triglide
Procedure: Cervical Conization — Cold knife conization or loop electrosurgical excision to remove cells and tissue in the cervix
  Arms: Excisional procedure + Fenofibrate
Procedure: Hysterectomy — In a hysterectomy, the uterus, cervix, both ovaries, both fallopian tubes, and nearby tissue are removed.
  Arms: Hysterectomy or chemoradiation + fenofibrate
Radiation: Chemoradiation — Chemotherapy uses anti cancer (cytotoxic) drugs to destroy cancer cells. The drugs circulate throughout the body in the bloodstream. Radiotherapy uses high energy waves similar to x-rays to kill cancer cells.
  Arms: Hysterectomy or chemoradiation + fenofibrate

SUMMARY:
Normally, p53 helps prevent tumors from forming in the body. Early studies have shown that Fenofibrate, a cholesterol-lowering drug, can restore normal function to p53 and can change the metabolism of HPV-positive tumors in a way that stops the growth of tumors. The purpose of this study is to understand how Fenofibrate can be used to treat HPV-positive cervical cancers and cervical dysplasia. Researchers will examine collected tissue samples and investigate various genes and proteins to see whether Fenofibrate has an effect on HPV-positive cervical cancers and cervical dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologic confirmed high grade dysplasia or cervical cancer. Histologic types include squamous cell, adenocarcinoma or adenosquamous cell carcinoma.
* Participants must be eligible for surgical management with LEEP, CKC or hysterectomy or chemoradiation
* Age ≥ 18 years
* Normal liver function (AST, ALT, bilirubin within institutional normal limits).
* Participants must be English speaking
* Participants must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with active liver disease, including primary biliary cirrhosis and unexplained, liver function abnormality
* Participants with severe kidney impairment (CrCl ≤30 mL/min calculated using Cockcroft-Gault), or end-stage kidney disease on dialysis
* Participants with preexisting gallbladder disease including active gallstones
* Known hypersensitivity to fenofibrate or fenofibric acid
* Participants that are pregnant or breast feeding due to unknown risk to developing fetus/infant. Please note: Participants of child-bearing potential (have had menses within the past year or have not had total hysterectomy) are actively screened for pregnancy prior to diagnostic procedures and screened again prior to treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in p53 levels | Up to six weeks after study enrollment
  Changes in p53 levels from initial biopsy to repeat sampling at the time of surgery
Change in tumor metabolic status | Up to six weeks after study enrollment
  Changes in tumor metabolic status from initial biopsy to repeat sampling at the time of surgery evaluated via immunohistochemical testing

SECONDARY OUTCOMES:
Fenofibrate tolerability | Up to six weeks after study enrollment
  Assess tolerability of fenofibrate by comparing lab values at baseline to values at conclusion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Ferguson, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States